CLINICAL TRIAL: NCT03709758
Title: Phase 1b Study of Venetoclax in Combination With Intensive Induction and Consolidation Chemotherapy in Treatment Naïve Subjects With Acute Myelogenous Leukemia
Brief Title: Venetoclax in Combination With Intensive Induction and Consolidation Chemotherapy in Treatment Naïve AML
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: AbbVie (Industry); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Richard Stone, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-351
Record Dates: First submitted 2018-10-12; First posted 2018-10-17 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Daunorubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Venetoclax+Daunorubicin+Cytarabine (Experimental): * Venetoclax administered orally on days 1 to 11 daily
  * Daunorubicin administered intravenously on days 2-4
  * Cytarabine administered on days 2-8 by continuous IV infusion
  Interventions: Drug: Venetoclax; Drug: Daunorubicin; Drug: Cytarabine

INTERVENTIONS:
Drug: Venetoclax — Venetoclax blocks an important pathway that promotes cell survival in tumor cells that overexpress BCL-2, so venetoclax causes cells to die
  Other Names: Venclexta
Drug: Daunorubicin — Chemotherapy is most effective at killing cells that are rapidly dividing.
  Other Names: Cerubidine
Drug: Cytarabine — Chemotherapy is most effective at killing cells that are rapidly dividing.
  Other Names: Cytosar-U

SUMMARY:
This research study is studying the combination of venetoclax and chemotherapy as a possible treatment for acute myelogenous leukemia (AML).

The drugs involved in this study are:

* Venetoclax
* Daunorubicin
* Cytarabine

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational drug and also tries to define the appropriate dose of the investigational drug to use for further studies. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved venetoclax for this specific disease but it has been approved for other uses.

In this research study, the investigators are combining the use of venetoclax (the investigational drug being studied) with chemotherapy drugs daunorubicin and cytarabine. The investigators are looking to determine the highest dose of venetoclax that can be given safely in combination with these chemotherapy drugs.

Depending on when the participant join the study, the participant may participate in part 1 (induction with venetoclax escalation), part 2 (consolidation with venetoclax escalation), or part 3 (an expansion cohort utilizing the maximum tolerated doses identified in parts 1 and 2). The study doctor will tell the participant which part of the study they will join.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML who are newly diagnosed according to the WHO 2016 Classification and previously untreated with the exception of hydroxyurea. ATRA pretreatment for suspected APL for less than 5 days is allowed. Eligible patients with AML arising from an antecedent hematologic disease (AHD) including MDS, may have been treated for their prior hematologic disease (except for allogenic transplant).
* AML patients include de-novo AML, AML evolving from MDS or other AHD and AML after previous cytotoxic therapy or radiation (secondary AML).

  * For a diagnosis of AML, a bone marrow or peripheral blast count of 20% or more is required.
  * In AML with monocytic or myelomonocytic differentiation, monoblasts and promonocytes, but not abnormal mature monocytes, are counted as blast equivalents.
* Patients must be ≥18 and ≤60 years old.
* Eastern Cooperative Oncology Group (ECOG) Performance status of 0 to 2. (See protocol Appendix D.)
* LVEF ≥ 45% by MUGA or ECHO at screening.
* Adequate renal function as demonstrated by a calculated creatinine clearance ≥ 50 mL/min; determined via urine collection for 24-hour creatinine clearance or by the Cockcroft Gault formula.
* Adequate liver function as demonstrated by:

  * aspartate aminotransferase (AST) ≤ 2.5 × ULN*
  * alanine aminotransferase (ALT) ≤ 2.5× ULN*
  * total bilirubin ≤ 1.5 × ULN*
* Unless considered due to leukemic organ involvement.
* Subjects with Gilbert's Syndrome may have a total bilirubin > 1.5 × ULN per discussion with the overall study PI
* Male subjects must agree to refrain from unprotected sex and sperm donation from initial study drug administration until 90 days after the last dose of study drug.
* Females of childbearing potential (i.e., not postmenopausal for at least 1 year or not surgically sterile) must have negative results by a serum pregnancy test performed within 7 days of day 1.
* Subject must voluntarily sign and date an informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria:

* Subject has acute promyelocytic leukemia, inversion16, t(8;21) or FLT3 mutant AML as described below. Contact PI with questions.

  * Inversion 16 and t(8;21): CBF chromosomal abnormalities may be assessed by molecular (PCR), metaphase cytogenetics, or FISH
  * FLT3: ITD or a point mutation in the TKD loop of variant allele fractions ≥5% by PCR, capillary electrophoresis, or NGS panel capable of defining FLT3 allelic burden
* Subject has known active CNS involvement with AML.
* Subject has tested positive for HIV (due to potential drug-drug interactions between antiretroviral medications and venetoclax, as well as anticipated venetoclax mechanism-based lymphopenia that may potentially increase the risk of opportunistic infections). Note: HIV testing is not required.
* Subject is known to be positive for hepatitis B or C infection with the exception of those with an undetectable viral load within 3 months. (Hepatitis B or C testing is not required). Subjects with serologic evidence of prior vaccination to HBV [i.e., HBs Ag-, and anti-HBs+] are allowed.
* Subject has received the following within 7 days prior to the initiation of study treatment:

  * Strong or moderate CYP3A inducers (see Appendix C)
  * Strong and moderate CYP3A inhibitors (see Appendix C)
* Subject has consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or Star fruit within 3 days prior to the initiation of study treatment.
* Subject has a cardiovascular disability status of New York Heart Association Class ≥ 2. Class 2 is defined as cardiac disease in which patients are comfortable at rest but ordinary physical activity results in fatigue, palpitations, dyspnea, or anginal pain.
* Subject has a significant history of renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, hepatic, cardiovascular disease, or any other medical condition that in the opinion of the investigator would adversely affect his/her participating in this study.
* Subject has chronic respiratory disease that requires continuous oxygen use.
* Subject has a malabsorption syndrome or other condition that precludes enteral route of administration.
* Subject exhibits evidence of other clinically significant uncontrolled condition(s) including, but not limited to: uncontrolled systemic infection.
* Subject has a history of other malignancies prior to study entry, with the exception of:

  * Adequately treated in situ carcinoma of the cervix uteri or carcinoma in situ of breast;
  * Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin;
  * Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent.
  * Prior malignancies treated with (surgery+/- chemotherapy+/- radiation) that have remained disease free for at least two years after completion of therapy
* Subject has a white blood cell count > 25 × 109/L. Note: Hydroxyurea is permitted to meet this criterion.
* Subject treated with any form of chemotherapy, immunotherapy, or investigative agent within 1 month of enrollment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2025-02-23 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (Induction) | 2 years
  To determine a safe and tolerable dose of venetoclax that can be given in combination with standard induction therapy to patients with newly diagnosed AML.
Maximum Tolerated Dose (Consolidation) | 2 years
  To determine a safe and tolerable dose of venetoclax and that can be given with a cycle of high dose cytarabine in consolidation after achievement of remission with induction therapy at the established MTD of venetoclax.

SECONDARY OUTCOMES:
Complete Response Rate | 2 years
  1. To obtain preliminary data as to the efficacy (Complete Remission (CR), Complete remission with incomplete platelet recovery (CRp), Complete remission with incomplete hematologic recovery (CRi), and minimal residual disease (MRD) negative CR) of combining venetoclax with standard induction and consolidation chemotherapy for AML.
Exploratory analysis concerning the impact of BH3 profiling on response when venetoclax is combined with standard induction and consolidation chemotherapy in AML. | 2 years
  BH3 profiling will be performed at the time of screening, and on PB blasts just prior to start of IV chemotherapy on day 2 of induction. These studies will determine if BH3 profile changes are induced by venetoclax exposure. Exploratory research analyses may not be included in the clinical study report.
Determine the pharmacodynamic effects of combo venetoclax with standard chemotherapy in AML on apoptosis and other intracellular events in AML blasts exposed in patients to a combination of venetoclax plus standard induction chemo. | 2 years
  A change in leukocytosis or blast counts will be evaluated as a measure of venetoclax-induced pharmacodynamic activity.
Exploratory analysis concerning the impact of pre-therapy disease factors including mutational profile on outcome in AML patients who receive venetoclax in combination with standard chemotherapy. | 2 years
  Single cell mass cytometry (CyTOF) will be used to observe changes in the levels of BCL-2 and associated proteins before therapy, at time of response assessment, upon recovery from consolidation (if applicable) and at relapse if feasible. Exploratory research analyses may not be included in the clinical study report.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Stone, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - University of Chicago, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No